CLINICAL TRIAL: NCT01746576
Title: Use of Near Infrared Spectroscopy to Measure Intracranial ScvO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Robert Thiele, MD, Assistant Professor, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16422
Record Dates: First submitted 2012-10-29; First posted 2012-12-11 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All (Other): All subjects will undergo spontaneous ventilation through an impedance threshold device and ScvO2 will be recorded before and after
  Interventions: Other: Use of impedance threshold device during spontaneous ventilation

INTERVENTIONS:
Other: Use of impedance threshold device during spontaneous ventilation

SUMMARY:
The purpose of this study is to determine whether analysis of near infrared absorbance signals that occur at different frequencies might provide information about the difference in oxygen saturation between arterial and venous blood.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18-65 years of age

Exclusion Criteria:

* Dilated cardiomyopathy
* Congestive heart failure
* Pulmonary hypertension
* Severe aortic stenosis
* Flail chest
* Chest pain
* Shortness of breath

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Estimated venous oxygen saturation | From 5 to 6:59 minutes after applying the impedance threshold device
  Oxygen saturation will be calculated from the five minute period of time prior to use of the impedance threshold device (0-4 mins), and then again in the 2 minute period after the impedance threshold device is applied (5-6 mins)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Thiele RH, Tucker-Schwartz JM, Lu Y, Gillies GT, Durieux ME. Transcutaneous regional venous oximetry: a feasibility study. Anesth Analg. 2011 Jun;112(6):1353-7. doi: 10.1213/ANE.0b013e3182166a26. PMID 21613200